CLINICAL TRIAL: NCT05577091
Title: Phase 1 Study of Autologous Tris-CAR-T Cell Locoregional Immunotherapy for Recurrent Glioblastoma
Brief Title: Tris-CAR-T Cell Therapy for Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Neurosurgical Institute (Other); Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Principal Investigator, Wei Zhang, Department of neurosurgery, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTSW2021-01
Record Dates: First submitted 2022-10-01; First posted 2022-10-13 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Glioblastoma
Keywords: Recurrent Glioblastoma; Immunotherapy; Adverse Events
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Recipients with the Ommaya reservoir implanted will be assigned to three courses. Arm A: Two patients, 1×10^7 autologous Tris-CAR-T, at least 1 dose, maximum 6 doses. Arm B: Two patients 1×10^8 autologous Tris-CAR-T, at least 1 dose, maximum 6 doses. Arm C: Six patients 5×10^7 autologous Tris-CAR-T, maximum 8 doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Tris-CAR-T cell (Experimental): Patients with supratentorial tumors for which CAR T cells will be delivered into the tumor resection cavity.
  Interventions: Genetic: Inverse correlated dual-target, truncated IL7Ra modified CAR -expressing autologous T-lymphocytes.

INTERVENTIONS:
Genetic: Inverse correlated dual-target, truncated IL7Ra modified CAR -expressing autologous T-lymphocytes. — Intratumoral or intraventricular administration via Ommaya reservoir.
  Dose level 0: 1×10^7 autologous Tris-CAR-T cells, at least one dose, maximum 6 doses, 2 patients.
  Dose level 1: 1×10^8/ 5×10^6 autologous Tris-CAR-T cells, at least one dose, maximum 6 doses, 2 patients. The dose of Dose level 1 will refer to the adverse effect of Dose level 0. When dose-related side effects occurred in 2 patients in the Dose level 0, the dose should be reduced to 5×10^6 cells.
  In Dose levels 0 and 1, the second dose will be infused 28 days after the first dose, and the subsequent doses will be administered weekly.
  Dose level 2: 5×10^7 autologous Tris-CAR-T cells, weekly administered, maximum 8 weeks, 4 patients. If the results of Dose levels 0 and 1 suggested that dose-related toxic side effects could have occurred in the 1×10^7cells dose, the researcher would re-determine the dosage of the multidose clinical exploration study.
  Other Names: Autologous Tris-CAR-T cell.

SUMMARY:
This is a Phase 1 study of recurrent glioblastoma locoregional adoptive therapy with autologous peripheral blood T cells lentivirally transduced to express a dual-target, truncated IL7Ra modified chimeric antigen receptor (CAR), delivered by Ommaya reservoir, a pre-indwelled catheter in the tumor resection cavity or ventricle. Patients with pathological confirmation of glioblastoma and radiological evidence of recurrence are candidates for this clinical trial. If the patient meets all other eligibility criteria, and meets none of the exclusion criteria, will have leukapheresis, and a subsequent Ommaya reservoir implantation. T cells will be isolated from the PBMC sample and then be bioengineered into a 4th generation CAR-T cell, Tris-CAR-T cells.

Recipients will be assigned to three courses in the order of enrollment. The first 2 patients will be assigned to the low-dose group. The second 2 patients will be assigned to the high dose group. The first 4 patients will have at least one dose of autologous Tris-CAR-T cells delivery via the Ommaya reservoir, at a maximum of 6 doses. The interval between the first and the second dose is 28 days, and the rest doses will be administered weekly. The last 6 patients will be assigned to the consecutive multidose group, and will receive a weekly dose of autologous Tris-CAR-T cells for a maximum of 8 weeks. All patients will undergo studies including MRI to evaluate the effect of the CAR-T cells, physical examination, and cerebrospinal fluid cytokine assays to evaluate side effects. All patients will undergo a long-term follow-up.

The hypothesis is that an adequate amount of Tris-CAR-T cells can be manufactured to complete all the three courses. The other hypothesis is that Tris-CAR-T cells can safely and effectively be administered through the Ommaya reservoir to allow the CAR-T cells to directly interact with the tumor cells for each patient enrolled in the study. The primary aim of the study will be to evaluate the safety of Tris-CAR-T administration. Secondary aims of the study will include evaluating CAR-T cell distribution within cerebrospinal fluid and peripheral blood, tumor progress post-CAR-T cell infusion, and, if tissue samples from multiple time points are available, also evaluate the degree of target expression, biological characteristics of samples at diagnosis versus at recurrence or progression.

DETAILED DESCRIPTION:
The autologous Tris-CAR-T cell, targeting both CD44 and CD133, the two inverse correlated targets, introduced truncated IL7Ra to the intracellular domain of the CAR molecule, and has shown ideal survival and tumor suppression in our previous studies. The cells will be tested for safety and kinetics in this clinical trial.

All patients are required to have an Ommaya reservoir in the tumor resection cavity before CAR-T cell infusion. Ommaya reservoir placement is done by surgery.

Autologous Tris-CAR-T cells will be manufactured via CliniMACS Instrument (Miltenyi Biotec). Cells will be thawed and sterily filled to infuse the patients. Each infusion will take between 5 and 10 minutes. We will then monitor the patient in the hospital for at least 3 days after the first dose of infusion. If the first infusion is tolerated well and the patient is assigned for multidose treatment, a second infusion may be given 28 days after the initial infusion for the first 4 patients (adverse effect assessment), and 7 days for the last 6 patients. Patients will be monitored in the hospital for no longer than 1 day. And the subsequent infusion will be done in the same manner. The treatment will be proceeded in the Department of Neurosurgery, Beijing Tiantan Hospital. Patients who receive multidose treatment will need to stay in Beijing for up to 8 weeks from the first infusion so we can monitor for side effects and will be readmitted to the hospital if patient develops a fever. If patient develops severe fevers after discharge from the hospital, the patient will be readmitted to the hospital for close monitoring for at least one night for safety observation and adverse effects management.

The first 4 patients will have follow-up visits at weeks 2, 3, and 4, then at months 3, 6, and 9 post-infusion. Patients of the consecutive multidose group will have follow-up visits at week 2, then at months 1 and 3 post-infusion. All patients receive long-term twice a year for a total of 15 years.

Medical tests before treatment--

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam
* Blood routine, serum biochemical test, kidney and liver function
* Measurements of the tumor by routine MRI

Medical tests during and after treatment--

The patient will receive standard medical tests when they are getting the infusions and afterward:

* Physical exams
* Blood routine, serum biochemical test, kidney and liver function, serum and (or) cerebrospinal fluid analysis
* Measurements of the tumor by MRI. Cerebrospinal fluid may be drawn from the patient's existing Ommaya reservoir preferentially, or via lumbar puncture before each infusion and at each time of follow-up. This procedure can be done at the bedside under local anesthesia and about 1ml of cerebrospinal fluid will be removed. Additional cerebrospinal fluid may be removed when intracranial hypertension occurs or other clinical needs.

To learn more about the pharmacokinetics of autologous Tris-CAR-T cells, peripheral blood will be obtained simultaneously with the cerebrospinal fluid collection. The amount of blood taken will be based on clinical need, for approximately 5 mL each time.

If the tumor samples of the patients are obtained, we will request a sample to be used for research purposes.

The patient will receive supportive care for any acute or chronic cytotoxicity, including blood components, cytokine antagonists, glucocorticoids, antibiotics, and other interventions as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years to 70 years (including cut-off values).
2. Patients with history of glioblastoma are diagnosed with recurrent glioblastoma and residual tumor after intracranial tumor resection/biopsy performed in Beijing Tiantan Hospital.
3. Patients who finished radiotherapy or temozolomide/bevacizumab or other drugs for at least 4 weeks. All toxicities of prior treatment should be defined as less than or equal to grade 1 (except for toxicities such as hair loss or leukoplakia) according to the Common Terminology Standard for Adverse Events (CTCAE 5.0).
4. Patients who is suitable for craniotocerebrospinal fluid shunt and attachment (Ommaya device) implantation confirmed by a competent physician.
5. Patients and/or legal representative is able to sign written informed consent.
6. Kanovsky Performance Status (KPS) ≥ 70.
7. According to the researchers' judgment, the life expectancy ≥ 8 weeks.
8. White blood cells (WBC) > 3.50×10^9/L (performed within 14 days prior to PBMC collection unless otherwise noted).
9. Platelet ≥ 200×10^9/L (performed within 14 days prior to PBMC collection unless otherwise noted).
10. Hemoglobin ≥ 120 g/L (performed within 14 days prior to PBMC collection unless otherwise noted).
11. Total bilirubin ≤ 20 μmol/L (performed within 14 days prior to PBMC collection unless otherwise noted).
12. Aspartic acid aminotransferase (AST) ≤ 2.5×42 U/L (performed within 14 days prior to PBMC collection unless otherwise noted).
13. Alanine aminotransferase (ALT) ≤ 2.5×41 U/L (performed within 14 days prior to PBMC collection unless otherwise noted).
14. Serum creatinine ≤ 90 μmol/L (performed within 14 days prior to PBMC collection unless otherwise noted).
15. Blood oxygen saturation ≥ 95% (performed within 14 days prior to PBMC collection unless otherwise noted).
16. Seronegative of the combination of human immunodeficiency virus (HIV) antibody (Ab) (performed within 14 days prior to PBMC collection unless otherwise noted).
17. Fertile women: a negative serum pregnancy test (performed within 14 days prior to PBMC collection unless otherwise noted).
18. The patient agrees that contraception should be used in patients of childbearing age for at least 3 months from screening to the last infusion of Tris-CAR-T cells. The period of childbearing age is defined as unsurgically neutered (men and women) or without menopause for more than 1 year (women only).

Exclusion Criteria:

1. Kanovsky Performance Status (KPS) ≤ 70.
2. Highly allergic constitution or severe allergies history.
3. Those who have psychiatric or psychological diseases and cannot cooperate with treatment and efficacy assessment.
4. Receive other drug trials within 60 days before enrollment, or receive other routine treatment in non-experimental designs for glioblastoma, such as stereotactic radiation therapy or placement of carmustine wafers.
5. Combined with infection, active infection, fever of unknown cause.
6. Combined with serious or unstable heart, lung, liver, kidney and hematopoietic system diseases, including active hepatitis.
7. Combined with inflammation and immune system diseases (such as rheumatoid arthritis), or known immunosuppressive diseases.
8. Combined with neurological diseases, such as diffuse leptomeningeal disease, or neurodegenerative diseases.
9. Known allergies to immunotherapy and related cellular products.
10. Patients who have received any gene therapy before.
11. Long-term use of immunosuppressants is required for any reason.
12. Patients with a history of organ transplantation or who are waiting for organ transplantation.
13. Special cases: pregnancy or lactation.
14. Other circumstances in which the investigators believe the patient is unsuitable for this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety: any adverse events associated with one or multiple autologous Tris-CAR-T cell infusions will be assessed by CTCAE v5.0. | 6 months
  Assesing the type, frequency, severity, and duration of adverse events as a result of autologous Tris-CAR-T cell infusion via physical, laboratory and imaging examination.

SECONDARY OUTCOMES:
CAR-T pharmacokinetics: the distribution, persistence of autologous Tris-CAR-T cell in the cerebrospinal fluid (CSF) and peripheral blood will be measured by qPCR. | 6 months
  The trafficking of autologous Tris-CAR-T cell in the CSF and peripheral blood will be assessed by quantifying the mRNA of CAR gene at the time of each infusion as well as at each time of follow-up via CSF extraction/ lumbar puncture and blood collection. CSF and peripheral blood will be collected prior to the initial infusion and will be set as baseline.
CAR-T pharmacodynamics: chemokines and cytokines produced by autologous Tris-CAR-T cell in the cerebrospinal fluid (CSF) and peripheral blood will be measured by Olink Proteomics. | 6 months
  The effect and its persistence of autologous Tris-CAR-T cell in the CSF and peripheral blood will be assessed via investigating the concentration of chemokines and cytokines. CSF and peripheral blood samples will be harvested at the time of each infusion as well as at each time of follow-up via CSF extraction/ lumbar puncture and blood collection. IL-6, TNF-α, IFN-γ, CCL2, CXCL10, G-CSF, GM-CSF, IL-10, IL-15, IL-7 and IL-1α will be investigated. CSF and peripheral blood will be collected prior to the initial infusion and will be set as baseline.
CAR-T therapeutic effect evaluation: the therapeutic effect of autologous Tris-CAR-T cell will be assessed by iRANO. | 12 months
  The total lesions will be mesured by MRI. Total lesions will be collected and calcultated prior to the initial infusion and will be set as baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Prof., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bagley SJ, Logun M, Fraietta JA, Wang X, Desai AS, Bagley LJ, Nabavizadeh A, Jarocha D, Martins R, Maloney E, Lledo L, Stein C, Marshall A, Leskowitz R, Jadlowsky JK, Christensen S, Oner BS, Plesa G, Brennan A, Gonzalez V, Chen F, Sun Y, Gladney W, Barrett D, Nasrallah MP, Hwang WT, Ming GL, Song H, Siegel DL, June CH, Hexner EO, Binder ZA, O'Rourke DM. Intrathecal bivalent CAR T cells targeting EGFR and IL13Ralpha2 in recurrent glioblastoma: phase 1 trial interim results. Nat Med. 2024 May;30(5):1320-1329. doi: 10.1038/s41591-024-02893-z. Epub 2024 Mar 13. PMID 38480922
- [Background] Choi BD, Gerstner ER, Frigault MJ, Leick MB, Mount CW, Balaj L, Nikiforow S, Carter BS, Curry WT, Gallagher K, Maus MV. Intraventricular CARv3-TEAM-E T Cells in Recurrent Glioblastoma. N Engl J Med. 2024 Apr 11;390(14):1290-1298. doi: 10.1056/NEJMoa2314390. Epub 2024 Mar 13. PMID 38477966
- [Background] Brown CE, Hibbard JC, Alizadeh D, Blanchard MS, Natri HM, Wang D, Ostberg JR, Aguilar B, Wagner JR, Paul JA, Starr R, Wong RA, Chen W, Shulkin N, Aftabizadeh M, Filippov A, Chaudhry A, Ressler JA, Kilpatrick J, Myers-McNamara P, Chen M, Wang LD, Rockne RC, Georges J, Portnow J, Barish ME, D'Apuzzo M, Banovich NE, Forman SJ, Badie B. Locoregional delivery of IL-13Ralpha2-targeting CAR-T cells in recurrent high-grade glioma: a phase 1 trial. Nat Med. 2024 Apr;30(4):1001-1012. doi: 10.1038/s41591-024-02875-1. Epub 2024 Mar 7. PMID 38454126
- [Background] Majzner RG, Ramakrishna S, Yeom KW, Patel S, Chinnasamy H, Schultz LM, Richards RM, Jiang L, Barsan V, Mancusi R, Geraghty AC, Good Z, Mochizuki AY, Gillespie SM, Toland AMS, Mahdi J, Reschke A, Nie EH, Chau IJ, Rotiroti MC, Mount CW, Baggott C, Mavroukakis S, Egeler E, Moon J, Erickson C, Green S, Kunicki M, Fujimoto M, Ehlinger Z, Reynolds W, Kurra S, Warren KE, Prabhu S, Vogel H, Rasmussen L, Cornell TT, Partap S, Fisher PG, Campen CJ, Filbin MG, Grant G, Sahaf B, Davis KL, Feldman SA, Mackall CL, Monje M. GD2-CAR T cell therapy for H3K27M-mutated diffuse midline gliomas. Nature. 2022 Mar;603(7903):934-941. doi: 10.1038/s41586-022-04489-4. Epub 2022 Feb 7. PMID 35130560
- [Background] Vitanza NA, Johnson AJ, Wilson AL, Brown C, Yokoyama JK, Kunkele A, Chang CA, Rawlings-Rhea S, Huang W, Seidel K, Albert CM, Pinto N, Gust J, Finn LS, Ojemann JG, Wright J, Orentas RJ, Baldwin M, Gardner RA, Jensen MC, Park JR. Locoregional infusion of HER2-specific CAR T cells in children and young adults with recurrent or refractory CNS tumors: an interim analysis. Nat Med. 2021 Sep;27(9):1544-1552. doi: 10.1038/s41591-021-01404-8. Epub 2021 Jul 12. PMID 34253928